CLINICAL TRIAL: NCT07278869
Title: Early Feasibility Study of the Append System for Left Atrial Appendage (LAA) Elimination by Invagination and Ligation
Brief Title: Applause Study I - Append System Early Feasibility Study
Acronym: Applause
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Append Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-000001
Record Dates: First submitted 2025-12-03; First posted 2025-12-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non Valvular Atrial Fibrillation
Keywords: Left Atrial Appendage (LAA)

STUDY DESIGN:
Intervention Model Description: Single-arm study in which all enrolled participants receive the Append System procedure
Masking Description: Not applicable - open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Append System (Experimental): Elimination of the left atrial appendage (LAA) using the Append System through a transcatheter procedure that invaginates and ligates the LAA tissue.
  Interventions: Device: Left Atrial Appendage Elimination: Append System

INTERVENTIONS:
Device: Left Atrial Appendage Elimination: Append System — Elimination of the left atrial appendage using the Append System through a transcatheter procedure involving invagination and ligation of the LAA tissue.

SUMMARY:
This early feasibility study is intended to evaluate the safety and feasibility of the Append System for eliminating the left atrial appendage (LAA) through a transcatheter procedure that invaginates and ligates the LAA tissue.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and performance of the Append System in patients with non-valvular atrial fibrillation who are considered appropriate candidates for LAA closure to reduce the risk of thromboembolism originating from the LAA.

The Append System is designed to eliminate the LAA without the use of a permanent metallic implant. The procedure is performed via a transfemoral, transseptal, transcatheter approach. During the procedure, the LAA is invaginated into the left atrium (LA), and the inverted tissue is ligated using a standard surgical suture, resulting in elimination of the LAA cavity.

Patients will be followed for up to 5 years after the procedure to assess safety, device performance, and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female aged ≥18 years
2. Documented non-valvular AF (paroxysmal, persistent, permanent or non-rheumatic valve-related AF)
3. The subject has a calculated CHA2DS2-VASc score of 2 or greater for males or 3 or greater for females.
4. The subject is eligible for the defined protocol medication regimen of anticoagulation and antiplatelet therapy following Append procedure.
5. The patient is deemed appropriate for LAA ligation by the screening committee and the investigator.
6. The patient has been informed of the nature of the study, agrees to its provisions & follow-up evaluations, and has provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC).

General Exclusion Criteria:

1. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following the index procedure. Female patients of childbearing potential must have a negative pregnancy test (per site standard test) within 7 days prior to index procedure.
2. Atrial fibrillation that is defined by a single occurrence or that is considered to be reversible (e.g., due to thyroid disorders, acute alcohol intoxication, trauma, or recent major surgical procedures).
3. Patients with an indication for chronic oral anticoagulation other than AF (e.g., history of unprovoked deep vein thrombosis or pulmonary embolism, or mechanical heart valve)
4. Clinically significant Severe heart failure (New York Heart Association functional class IV)
5. Prior cardiac surgery or surgery requiring sternotomy
6. Recent (within 3 months pre-procedure) stroke or transient ischemic attack.
7. Recent (within 3 months pre-procedure) myocardial infarction
8. Recent (within 30 days before the index procedure) or planned (within 60 days after the index procedure) cardiac interventional procedures (e.g., percutaneous coronary intervention, structural heart valve procedures, etc.)
9. Planned (within 60 days after the index procedure) cardiac surgical procedures or any surgeries which require sternotomy.
10. Recent (within 30 days before the index procedure) or planned (within 60 days after the index procedure) noncardiac procedures or surgical interventions.
11. History of symptomatic pericarditis (acute or chronic).
12. Patient has evidence of cardiac tumor
13. Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 (by the Modification of Diet in Renal Disease equation), or dialysis at the time of screening
14. Platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <3,000 cells/mm3 or known Bleeding diathesis
15. Active infection with bacteremia
16. Patient has a known allergy, hypersensitivity or contraindication to aspirin, heparin, or that would preclude any P2Y12 inhibitor therapy, or the patient has contrast sensitivity that cannot be adequately pre-medicated
17. Current participation in another investigational drug or device study that would interfere with this study
18. Patient is unable to undergo general anesthesia
19. Patient has a condition which precludes adequate transesophageal echocardiographic (TEE) or computed tomographic (CT) assessment.
20. Known other medical illness or known history of substance abuse that may cause non-compliance with the specified medication regimen, confound the data interpretation, or is associated with a life expectancy of less than 5 years.

Cardiac Imaging Exclusion Criteria:

1. Intracardiac thrombus observed during screening
2. Left ventricular ejection fraction (LVEF) <30%
3. Circumferential pericardial effusion >5 mm or signs / symptoms of acute or chronic pericarditis, or evidence of tamponade physiology
4. Distance from inter-atrial septum fossa ovalis to LAA ostium is less than 40 mm
5. Any anatomy or prior intervention that would preclude a transseptal approach (including, but not limited to, prior IVC filter placement that cannot be crossed, prior ASD, or prior PFO closure device implantation that precludes transseptal puncture)
6. LAA structure that in the opinion of the screening committee / investigator precludes intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Composite major adverse events | 30 days
  Composite rate of major adverse events related to the device or procedure, including all-cause mortality, ischemic stroke, systemic embolism, and cardiac tamponade or pericardial effusion requiring drainage

SECONDARY OUTCOMES:
Composite major adverse events | 6 months
  Composite rate of major adverse events related to the device or procedure, including all-cause mortality, ischemic stroke, systemic embolism, pericardial effusion requiring drainage, major bleeding (BARC 3/ BARC 5), hemorrhagic stroke, and device or procedure-related events requiring open cardiac surgery or major endovascular intervention such as pseudoaneurysm repair, AV fistula repair, or other major endovascular repair
Procedure and Technical Success | 30 days
  LAA cavity elimination by LAA invagination and ligation with invagination proximal to the LAA ostium and lack of fluid communication between the LA and LAA- observed by TEE

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The study is an early feasibility investigation conducted under an FDA IDE, and the data will be retained by the sponsor and reported in aggregate only.